CLINICAL TRIAL: NCT02672046
Title: Danish Title: Optimeret Visitation af Midaldrende knæpatienter Med Symptomer Muligvis Relateret Til Meniskskade
Brief Title: Optimized Referral of Knee Patients at the Clinic of Sports Injuries
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 6300002
Record Dates: First submitted 2016-01-20; First posted 2016-02-03 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2016-01

CONDITIONS: Knee Injuries; Knee; Injury, Meniscus (Lateral) (Medial)
MeSH Terms: conditions — Knee Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with knee injuries: Patients referred to assessment at the Clinic of Sports Injuries
  Interventions: Other: Assessment at the Clinic of Sports Injuries

INTERVENTIONS:
Other: Assessment at the Clinic of Sports Injuries — Assessment at the Clinic of Sports Injuries as well as a new algorithm (using patient-reported symptoms will be applied

SUMMARY:
The aim of the study is to evaluate an algorithm to screen patients with a possibility of meniscal injury referred to a sports injury outpatient clinic by using patient-reported symptoms. It will be investigated whether the algorithm is able to identify which patients are deemed relevant to undergo assessment by a physician (i.e. in case the patient need to undergo surgery) and which patients are relevant to undergo assessment by a physiotherapist. This will be evaluated by estimating the sensitivity of the new algorithm compared to actual relevancy based on the traditional clinical assessment of the patients.

DETAILED DESCRIPTION:
According to current practice, patients referred to the Clinic of Sports Injuries will be assessed by either a physician or a physiotherapist. Current practice will continue unchanged during this study.

Before the scheduled assessment, patients will be asked to fulfill a questionnaire including KOOS, a further description of symptoms, previous treatment by physiotherapist and expected upcoming treatment (i.e. surgery or referral to physiotherapist).

An algorithm based on the self-reported information will be used to categorize whether the patient are considered relevant to be referred to assessment by a physician or to assessment by a physiotherapist.

After clinical assessment of the patient, the physician or physiotherapist does a registration of diagnosis, choice of treatment and complexity. Based on choice of treatment and complexity, the patient will be categorized as either relevant to be referred to assessment by a physician or to assessment by a physiotherapist. This categorization is by definition considered correct.

The ability of the algorithm will be evaluated by comparing it's categorization to the correct result. Sensitivity will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 35 referred to the Clinic of Sports Injuries with knee symptoms

Exclusion Criteria:

* Cognitive or language problems that precludes the filling of the questionnaires
* Previous surgery in the knee
* Symptoms only located in the anterior part of the knee

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Middle aged patients with knee symptoms referred to the Clinic of Sports Injuries
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
"Relevant referral to assessment by physician" or "Relevant referral to assessment by physiotherapist" | Up to 4 weeks (at the initial visit at the Clinic of Sports Injuries)

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At baseline

OTHER OUTCOMES:
Choice of treatment | Up to 4 weeks (at the initial visit at the Clinic of Sports Injuries)
  Referral to physical therapy, surgery, information and advice, other

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nørgaard Madsen, PT, Principal Investigator — University of Aarhus
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No